CLINICAL TRIAL: NCT01895101
Title: The Effect on Blood Loss of Topical and Intravenous Tranexamic Acid in Cardiac Surgery Patients: a Randomized Placebo-controlled Trial
Brief Title: The Effect on Blood Loss of Topical and Intravenous Tranexamic Acid in Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Thierry V Scohy, MD, phd, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-1251; 2013-000774-30 (EudraCT Number)
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Blood Loss; Tranexamic Acid; Cardiac Surgery
Keywords: blood loss; tranexamix acid; cardiac surgery
MeSH Terms: conditions — Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pericardial lavage with 200 ml normothermic saline solution (Placebo Comparator): According to the anaesthetic protocol of the Amphia Hospital (Breda, the Netherlands), all patients scheduled for cardiac surgery receive intravenously 2 gr TA before sternal incision and 2 gr TA after cardiopulmonary bypass.
  This arm also receives pericardial lavage with 200 ml normothermic saline solution without tranexamic acid.
  Interventions: Drug: Saline
- No pericardial lavage (No Intervention): According to the anaesthetic protocol of the Amphia Hospital (Breda, the Netherlands), all patients scheduled for cardiac surgery receive intravenously 2 gr TA before sternal incision and 2 gr TA after cardiopulmonary bypass.
  In this arm the subjects receives as in standard care no pericardial lavage.
- 2 gr tranexamic acid diluted in 200 ml normothermic saline (Experimental): According to the anaesthetic protocol of the Amphia Hospital (Breda, the Netherlands), all patients scheduled for cardiac surgery receive intravenously 2 gr TA before sternal incision and 2 gr TA after cardiopulmonary bypass.
  This arm receives also pericardial lavage with 2 gr TA diluted in 200 ml normothermic saline solution (NaCl 0.9%).
  Interventions: Drug: 2 gr tranexamic acid

INTERVENTIONS:
Drug: 2 gr tranexamic acid — This group receives pericardial lavage with 2 gr tranexamic diluted in 200 ml normothermic saline solution (NaCl 0.9%).
  Arms: 2 gr tranexamic acid diluted in 200 ml normothermic saline
Drug: Saline — This group receives pericardial lavage with 200 ml normothermic saline solution without tranexamic acid
  Arms: pericardial lavage with 200 ml normothermic saline solution

SUMMARY:
It remains still unclear whether topical tranexamic acid has an added value besides the administration of intravenously tranexamic acid. We hypothesize that the addition of topical tranexamic acid, besides intravenous administration of tranexamic acid, results in a 25% reduction of post-operative blood loss after cardiac surgery.

The aim of this study is to determine whether the application of topical tranexamic acid reduces the 12 hours postoperative blood loss by 25% in patient scheduled for cardiac surgery on cardiopulmonary bypass, whereby intravenous tranexamic acid is administrated.

Just before sternal closure, 250 subjects receives pericardial lavage with 2 gr tranexamic acid in 200 ml normothermic saline solution (NaCl 0.9%), 250 subjects receives pericardial lavage with 200 ml normothermic saline solution without TA and 250 subjects (control group) receives no pericardial lavage. The main study parameter is 12 hours post-operative blood loss and is assessed by 12 hours post-operative chest tube production.

ELIGIBILITY:
Inclusion Criteria:

* Gender; male/ female
* Age: ≥ 18 year
* Elective cardiac surgical patients

  * Coronary artery bypass graft (CABG) (conventional, E.CCO)
  * Aortic valve replacement (AVR) (conventional)
  * Mitral valve replacement (MVR)/ Mitral valve repairment (MPL) (conventional)
  * Tricuspid valve replacement (TVR) / Tricuspid valve repairment (TPL)
  * Bentall
  * Combined procedure (e.g. CABG/ AVR, MVR/AVR, AVR/Maze)

Exclusion Criteria:

* MVR/MPL (minimal invasive, Port Access Surgery)
* Maze (minimal invasive, via Thoracoscopy)
* AVR (minimal invasive, via mini Sternotomy)
* off-pump procedures
* Emergency operations
* Patient with increased or decreased blooding tendency (FV leiden, prot C, S deficiency, anti-thrombin deficiency, prothrombin mutation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Scohy, Principal Investigator — Amphia Hospital
Locations (1):
- Amphia Hospital, Breda, Netherlands

REFERENCES:
- [Background] Mahaffey R, Wang L, Hamilton A, Phelan R, Arellano R. A retrospective analysis of blood loss with combined topical and intravenous tranexamic acid after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2013 Feb;27(1):18-22. doi: 10.1053/j.jvca.2012.08.004. Epub 2012 Oct 10. PMID 23063104
- [Background] De Bonis M, Cavaliere F, Alessandrini F, Lapenna E, Santarelli F, Moscato U, Schiavello R, Possati GF. Topical use of tranexamic acid in coronary artery bypass operations: a double-blind, prospective, randomized, placebo-controlled study. J Thorac Cardiovasc Surg. 2000 Mar;119(3):575-80. doi: 10.1016/s0022-5223(00)70139-5. PMID 10694619
- [Background] Baric D, Biocina B, Unic D, Sutlic Z, Rudez I, Vrca VB, Brkic K, Ivkovic M. Topical use of antifibrinolytic agents reduces postoperative bleeding: a double-blind, prospective, randomized study. Eur J Cardiothorac Surg. 2007 Mar;31(3):366-71; discussion 371. doi: 10.1016/j.ejcts.2006.12.003. Epub 2007 Jan 10. PMID 17218108
- [Background] Abul-Azm A, Abdullah KM. Effect of topical tranexamic acid in open heart surgery. Eur J Anaesthesiol. 2006 May;23(5):380-4. doi: 10.1017/S0265021505001894. Epub 2006 Jan 27. PMID 16438759
- [Background] Spegar J, Vanek T, Snircova J, Fajt R, Straka Z, Pazderkova P, Maly M. Local and systemic application of tranexamic acid in heart valve surgery: a prospective, randomized, double blind LOST study. J Thromb Thrombolysis. 2011 Oct;32(3):303-10. doi: 10.1007/s11239-011-0608-3. PMID 21660523

RESULTS

PARTICIPANT FLOW:
Groups:
- Pericardial Lavage With 200 ml Normothermic Saline Solution: According to the anaesthetic protocol of the Amphia Hospital (Breda, the Netherlands), all patients scheduled for cardiac surgery receive intravenously 2 gr TA before sternal incision and 2 gr TA after cardiopulmonary bypass.
  This arm also receives pericardial lavage with 200 ml normothermic saline solution without tranexamic acid.
  Saline: This group receives pericardial lavage with 200 ml normothermic saline solution without tranexamic acid
- 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline: According to the anaesthetic protocol of the Amphia Hospital (Breda, the Netherlands), all patients scheduled for cardiac surgery receive intravenously 2 gr TA before sternal incision and 2 gr TA after cardiopulmonary bypass.
  This arm receives also pericardial lavage with 2 gr TA diluted in 200 ml normothermic saline solution (NaCl 0.9%).
  2 gr tranexamic acid: This group receives pericardial lavage with 2 gr tranexamic diluted in 200 ml normothermic saline solution (NaCl 0.9%).
Period: Overall Study
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline
Started | 250 | 250 | 250
Completed | 249 | 245 | 245
Not Completed | 1 | 5 | 5
Not completed — OPCAB procedure | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — another study, enrolled in other study | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — coagulation disorder | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline | Total
Number analyzed (Participants) | 249 | 245 | 245 | 739
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [62 to 75] | 68 [63 to 76] | 69 [62 to 75] | 69 [62 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 65 | 49 | 159
  Male | 204 | 180 | 196 | 580
Region of Enrollment [Number; unit: participants]
  Netherlands | 249 | 245 | 245 | 739

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Blood Loss
Description: The primary study parameter is 12 hours postoperative blood loss and is assessed by postoperative chest tube production. Postoperative chest tube production 12 hours after surgical procedure
Time Frame: 12 hours postoperative
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline
Number analyzed (Participants) | 249 | 245 | 245
ml | 290 [210 to 410] | 300 [190 to 450] | 290 [190 to 430]

2. Secondary Outcome: Number of Participants Requiring Surgical Re-exploration
Description: the secondary objective of this study is to determine whether pericardial lavage with saline gives an improvement in haemostasis, compared with no pericardial lavage, resulting in a reduction of surgical re-explorations and post-operative 12-hour blood loss. The choice for a surgical re-exploration will be decided according to the ICU protocol.
Time Frame: participants will be followed for the duration of ICU stay, an expected average of 2 days
Measure: Number; unit: participants
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline
Number analyzed (Participants) | 249 | 245 | 245
participants | 10 | 9 | 12

3. Secondary Outcome: Total Red Blood Cell Transfusions (Cumulative of Pre, Peri and Postoperative Period)
Description: The amount of red blood cell transfusions the patient receive pre, peri and postoperatively during their stay in the hospital.
Time Frame: participants will be followed for the duration of ICU stay, an expected average of 2 days/ And participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline
Number analyzed (Participants) | 249 | 245 | 245
IU | 0.7 (1.6) | 1.1 (3.2) | 0.7 (1.5)

ADVERSE EVENTS:
Arm/Group | Pericardial Lavage With 200 ml Normothermic Saline Solution | No Pericardial Lavage | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline
Serious Adverse Events (participants affected / at risk) | 7/250 | 4/250 | 4/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250 | 0/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pericardial Lavage With 200 ml Normothermic Saline Solution (N=250) | No Pericardial Lavage (N=250) | 2 gr Tranexamic Acid Diluted in 200 ml Normothermic Saline (N=250)
cerebrovascular accident (General disorders) | 3 | 1 | 2
Death (Cardiac disorders) | 4 | 2 | 2
epileptic seizures (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes